CLINICAL TRIAL: NCT00309556
Title: A Randomized Phase III Study Comparing Epirubicin, Docetaxel and Capecitabine + G-CSF to Epirubicin and Docetaxel + G-CSF as Neoadjuvant Treatment for Early HER-2 Negative Breast Cancer and Comparing Epirubicin, Docetaxel and Capecitabine + G-CSF ± Trastuzumab to Epirubicin and Docetaxel + G-CSF ± Trastuzumab as Neoadjuvant Treatment for Early HER-2 Positive Breast Cancer
Brief Title: Randomized Neoadjuvant Study of Epirubicin and Docetaxel With/Without Capecitabine in Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Amgen (Industry); Ebewe Pharma GmbH (Unknown); Hoffmann-La Roche (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG-24; Ro 09-1978 (Other: Roche Study ID)
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: Epirubicin; Docetaxel; Capecitabine; Herceptin; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Docetaxel; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (experimental group) (Active Comparator): Epirubicin/Docetaxel/Capecitabine-containing chemotherapy ± trastuzumab in HER-2 positive disease
  Interventions: Drug: Epirubicin; Drug: Docetaxel; Drug: Capecitabine; Drug: Trastuzumab
- B (control group) (Active Comparator): Epirubicin/Docetaxel-containing chemotherapy ± trastuzumab in HER-2 positive disease
  Interventions: Drug: Epirubicin; Drug: Docetaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Epirubicin — 6 cycles 75mg/m2 i.v. day 1 q3w
Drug: Docetaxel — 6 cycles 75mg/m2 i.v. day 1 q3w
  Other Names: Taxotere
Drug: Capecitabine — 6 cycles 1000mg/m2 oral, day 1-14 q2d
  Other Names: Xeloda
  Arms: A (experimental group)
Drug: Trastuzumab — cycle 1: 8mg/kg i.v. day 1 cycle 2-6: 6mg/kg i.v. day 1 (=6 cycles q3w)
  Other Names: Herceptin

SUMMARY:
Primarily, this clinical investigation compares the rates (percentages) of pathological complete remissions attained at the time of final surgery following 6 cycles each of epirubicin + docetaxel + capecitabine-containing chemotherapy ± trastuzumab (in HER-2 positive disease) vs. epirubicin + docetaxel-containing chemotherapy ± trastuzumab (in HER-2 negative disease).

DETAILED DESCRIPTION:
This study is a prospective, randomized, multicentre, phase III trial in the neoadjuvant treatment of patients with primary breast cancer and no distant metastases. Patients will be stratified at inclusion according to the centre, to the clinical tumour stage (T1, T2, T3, T4a-c), the axillary lymph node status (positive, negative), the menopausal status (pre-menopausal, post-menopausal), histology (invasive ductal, invasive lobular, mixed), the hormone-receptor status (positive [ER+/PR+, ER+/PR-, ER-/PR+], negative [ER-/PR-], not determinable]), the HER-2 status (positive, negative, not determinable), the grading (G1/G2, G3, not determinable) and will be randomly assigned to receive either 6 cycles of neoadjuvant epirubicin, docetaxel and capecitabine ± trastuzumab in HER-2 positive disease or 6 cycles of neoadjuvant epirubicin and docetaxel ± trastuzumab in HER-2 positive disease.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically proven, core-biopsied, invasive breast cancer of any clinical and/or radiological T-stage (except for T4d)
* Age 18-70 years
* WHO performance status ≤ 2
* No prior or current neoplasm except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix
* No distant disease / secondary carcinoma judged clinically and at least by chest X-ray, liver sonography, and bone scan upon randomization
* No medical and/or cardiologic contraindication to receive an anthracycline- and taxane-containing chemotherapy regimen. Normal cardiac function must be confirmed by LVEF (echocardiography or Muga scan). The result must be above 50% or above the institution's ULN
* Results of the following assessments at the time of randomization must be available:

  1. chest wall CT, abdomen CT, bilateral mammography: within 4 weeks before enrolment;
  2. laboratory requirements: within 2 weeks before enrolment
  3. hematology: neutrophils ≥ 4.0 x 109/l, platelets ≥ 150 x 109/l, haemoglobin ≥ 13 g/dl
  4. hepatic function: total bilirubin < 1 x ULN, ASAT (SGOT) and ALAT (SGPT) < 1x ULN, alkaline phosphatase < 1 x ULN. In case of abnormal values, liver function tests have to be repeated within 3 days before study treatment.
  5. renal function: creatinine ≤ 1 x ULN,
  6. histology, grading, hormone receptor status, HER-2/neu status
* Signed and dated informed consent before the start of specific protocol procedures
* Negative pregnancy test in the presence of childbearing potential

Exclusion Criteria:

* Stage T4d / inflammatory breast cancer
* Pregnant or lactating patients; patients of childbearing potential must implement adequate contraceptive measures during study participation
* Pre-existing motor or sensory neurotoxicity of a severity ≥ WHO grade 2
* Preoperative local treatment for breast cancer (i.e. incomplete surgery, radiotherapy)
* Prior or concomitant systemic antitumor therapy
* Other serious illness or medical condition

  1. congestive heart failure or unstable angina pectoris, even if medically controlled.

     Previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or high-risk uncontrolled arrythmias
  2. history of significant neurologic or psychiatric disorders, including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
  3. active uncontrolled infection
  4. unstable peptic ulcer, unstable diabetes mellitus or other contraindication for the use of corticosteroids
* Concurrent treatment with corticosteroids except as use for the prophylactic regimen, inhalational use, treatment of acute hypersensitivity reactions, treatment of nausea/vomiting or chronic treatment (initiated > 6 months prior to study entry) at low dose (≤ 20 mg methylprednisolone or equivalent)
* Known hypersensitivity against taxanes and/or epirubicin and/or fluorouracil/capecitabine
* Known dihydropyrimidine-dehydrogenase (DPD) deficit
* Treatment with an investigational drug within 30 days prior to study entry
* Legally incapacitated and/or other circumstances which make it unfeasible for the subject to understand the nature, meaning and consequences of the clinical study
* Concurrent psychiatric illness according to ICD (alcohol addiction) at the time of study entry

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2005-02; Primary Completion 2009-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Rate of pathological complete remissions | 20 weeks
  at the time of final surgery after 6 cycles of Arm A (Epirubicin/ Docetaxel/ Capecitabine-containing chemotherapy ± Trastuzumab in HER-2 positive disease) vs. Arm B (Epirubicin/Docetaxel-containing chemotherapy ± Trastuzumab in HER-2 positive disease).

SECONDARY OUTCOMES:
Rates of axillary lymph node involvement and breast-conserving procedures | 20 weeks
  at the time of final surgery in Arm A (± trastuzumab in HER-2 positive disease) vs. Arm B (± trastuzumab in HER-2 positive disease).

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Steger, MD, Study Chair — Austrian Breast & Colorectal Cancer Study Group
Locations (26):
- Austria (26):
  - Hospital Guessing, Güssing, Burgenland
  - Hospital Oberpullendorf, Oberpullendorf, Burgenland
  - Hospital Oberwart, Oberwart, Burgenland
  - State Hospital Klagenfurt, Klagenfurt, Carinthia
  - Ordination Dr. Wette, Saint Veit A. D. Glan, Carinthia
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit A. D. Glan, Carinthia
  - State Hospital Villach, Villach, Carinthia
  - State Hospital Wolfsberg, Wolfsberg, Carinthia
  - Hospital Baden, Baden, Lower Austria
  - Hospital Krems, Krems, Lower Austria
  - Hospital of Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Paracelsus Medical University Salzburg - Oncology, Salzburg, Salzburg
  - Gynaegological Medical University Graz, Graz, Styria
  - Medical University of Graz, Oncology, Graz, Styria
  - State Hospital Leoben, Leoben, Styria
  - Medical University of Innsbruck, Innsbruck, Tyrol
  - District Hospital Kufstein, Kufstein, Tyrol
  - State Hospital Kirchdorf, Kirchdorf, Upper Austria
  - Hospital BHS Linz, Linz, Upper Austria
  - General Hospital Linz, Linz, Upper Austria
  - State Hospital Steyr, Steyr, Upper Austria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - Medical University Vienna, General Hospital, Vienna, Vienna
  - State Hospital Vienna-Hietzing, Vienna, Vienna
  - Hanusch Hospital, Vienna, Vienna
  - State Hospital Feldkirch/Rankweil, Rankweil, Vorarlberg

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Steger GG, Greil R, Lang A, Rudas M, Fitzal F, Mlineritsch B, Hartmann BL, Bartsch R, Melbinger E, Hubalek M, Stoeger H, Dubsky P, Ressler S, Petzer AL, Singer CF, Muss C, Jakesz R, Gampenrieder SP, Zielinski CC, Fesl C, Gnant M; Austrian Breast and Colorectal Study Group (ABCSG). Epirubicin and docetaxel with or without capecitabine as neoadjuvant treatment for early breast cancer: final results of a randomized phase III study (ABCSG-24). Ann Oncol. 2014 Feb;25(2):366-71. doi: 10.1093/annonc/mdt508. Epub 2013 Dec 16. PMID 24347519
- See also: Click here for more information about this study: ABCSG-Studien closed — http://www.abcsg.at